CLINICAL TRIAL: NCT03364088
Title: Outcome After Total Knee Arthroplasty Under General or Spinal Anesthesia, a Randomized Controlled Trial
Brief Title: Outcome After Total Knee Arthroplasty Under General or Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riku Antero Palanne (Other)
Collaborators: Helsinki University Central Hospital (Other); University of Helsinki (Other); Finland (Unknown)
Responsible Party: Sponsor-Investigator, Riku Antero Palanne, Principal investigator, Helsinki University Central Hospital
Organization: Helsinki University Central Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PeijasTKA
Record Dates: First submitted 2017-10-30; First posted 2017-12-06 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Knee Osteoarthritis; Arthropathy of Knee Joint; Knee Pain Chronic; Rheumatoid Arthritis; Anesthesia
Keywords: Total knee arthroplasty; Anesthesia; Surgical tourniquet; Pain; Postoperative nausea and vomiting; Quality of life; Length of stay; Knee function; Bioelectrical impedance; Knee endoprosthesis
MeSH Terms: conditions — Osteoarthritis, Knee; Arthritis, Rheumatoid; Pain; Postoperative Nausea and Vomiting | interventions — Anesthesia, Spinal; Tourniquets; Anesthesia, General

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Spinal anesthesia with tourniquet (Active Comparator): This group will be operated under spinal anesthesia (15 mg of bupivacaine) and in continuous light propofol sedation. Surgical tourniquet (with the pressure of 250 mmHg or > 100 mmHg higher than systolic blood pressure) is used during the operation.
  Local infiltration analgesia (LIA) will be administered during the operation. Patients receive 1 g of intravenous tranexamic acid approximately 5 - 10 minutes before the removal of the tourniquet.
  Postoperatively patient-controlled analgesia (PCA) with intravenous oxycodone will be used for 24 hours.
  Interventions: Procedure: Spinal anesthesia with tourniquet; Drug: Oxycodone by patient-controlled analgesia (PCA)
- Spinal anesthesia without tourniquet (Active Comparator): This group will be operated under spinal anesthesia (15 mg of bupivacaine) and in continuous light propofol sedation. Surgical tourniquet is not used during the operation.
  Patients receive 1 g of intravenous tranexamic acid approximately 5 - 10 minutes before the surgical incision. Local infiltration analgesia (LIA) will be administered during the operation.
  Postoperatively patient-controlled analgesia (PCA) with intravenous oxycodone will be used for 24 hours.
  Interventions: Procedure: Spinal anesthesia without tourniquet; Drug: Oxycodone by patient-controlled analgesia (PCA)
- General anesthesia with tourniquet (Active Comparator): This group will be operated under general anesthesia (propofol and remifentanil are used with target-controlled infusion (TCI) mode) and surgical tourniquet (with the pressure of 250 mmHg or > 100 mmHg higher than systolic blood pressure) is used during the operation.
  Local infiltration analgesia (LIA) will be administered during the operation. Patients receive 1 g of intravenous tranexamic acid approximately 5 - 10 minutes before the removal of tourniquet. Intravenous bolus of oxycodone 0.1 mg/kg (ideal body weight) is given when the closure of surgical wound begins.
  Postoperatively patient-controlled analgesia (PCA) with intravenous oxycodone will be used for 24 hours.
  Interventions: Procedure: General anesthesia with tourniquet; Drug: Oxycodone by patient-controlled analgesia (PCA)
- General anesthesia without tourniquet (Active Comparator): This group will be operated under general anesthesia (propofol and remifentanil are used with target-controlled infusion (TCI) mode) without the use of surgical tourniquet.
  Patients receive 1 g of intravenous tranexamic acid approximately 5 - 10 minutes before the surgical incision. Local infiltration analgesia (LIA) will be administered during the operation. Intravenous bolus of oxycodone 0.1 mg/kg (ideal body weight) is given when the closure of surgical wound begins.
  Postoperatively patient-controlled analgesia (PCA) with intravenous oxycodone will be used for 24 hours.
  Interventions: Procedure: General anesthesia without tourniquet; Drug: Oxycodone by patient-controlled analgesia (PCA)

INTERVENTIONS:
Procedure: Spinal anesthesia with tourniquet — Operation is done under spinal anesthesia and surgical tourniquet is used.
  Arms: Spinal anesthesia with tourniquet
Procedure: Spinal anesthesia without tourniquet — Operation is done under spinal anesthesia and without the use of surgical tourniquet.
  Arms: Spinal anesthesia without tourniquet
Procedure: General anesthesia with tourniquet — Operation is done under general anesthesia and surgical tourniquet is used.
  Arms: General anesthesia with tourniquet
Procedure: General anesthesia without tourniquet — Operation is done under general anesthesia and without the use of surgical tourniquet.
  Arms: General anesthesia without tourniquet
Drug: Oxycodone by patient-controlled analgesia (PCA) — PCA device (CADD Legacy PCA Pump, Smiths Medical, Kent, UK) is programmed to give intravenous oxycodone in doses of 0.04 mg/kg (ideal body weight). The minimum time between doses is set to 10 minutes and no more than 4 doses per hour are allowed.

SUMMARY:
Previous retrospective database studies suggest that total knee arthroplasty (TKA) surgery under spinal anesthesia has less complications than when performed under general anesthesia. In general, complications are rare and both anesthesia types are widely accepted. In Finland, total knee arthroplasty has typically been performed under spinal anesthesia.

In a recent prospective randomized controlled study, total knee arthroplasty under general anesthesia resulted in less acute postoperative pain (opioid-need measured by patient-controlled anesthesia), less nausea, and faster hospital discharge than that performed under spinal anesthesia. Also the use of surgical tourniquet can affect surgical outcome: it may reduce bleeding and surgery time, but it may also cause weakness of thigh muscles and thus hinder mobilization. In a recent study, both techniques with and without surgical tourniquet appeared equal.

The aims of this study are to compare total knee arthroplasty under spinal or general anesthesia, with or without surgical tourniquet, in relation to acute and chronic postoperative pain, nausea, knee function, patient reported quality of life and satisfaction on care, complications, length of stay, and need of surgical unit resources. This randomized controlled study includes 400 patients with informed consent, 18-75-years-of-age, standard primary total knee arthroplasty operation, American Society of Anesthesiologist (ASA) physical status classification I-III, body mass index under 40, and no contraindications for medications or treatments used.

The hypothesis of this study are used to reassess best practices of primary total knee arthroplasty operation to enhance quality of care, patient outcomes and satisfaction, and availability of surgery due to better patient flow at surgical unit.

ELIGIBILITY:
Inclusion Criteria:

* Indication for total knee arthroplasty exists (patient has osteoarthritis, rheumatoid arthritis or other disease affecting knee joint that does not respond to conservative treatment)
* Patient understands the study information and is willing to participate
* Triathlon endoprosthesis is suitable for patient
* ASA Physical Status Classification 1-3
* Patient will be operated by a surgeon who has done at least 100 total knee arthroplasty procedures with Triathlon endoprosthesis before

Exclusion Criteria:

* BMI > 40 kg/m2
* ASA Physical Status Classification > 3
* Valgus or varus > 15° degrees in the knee that will be operated
* Extension deficit ≥ 20° or flexion ≤ 90° in the knee that will be operated
* Earlier major (open) surgery in the knee that will be operated
* Contraindication for drugs used in the study
* Contraindication for either spinal or general anesthesia
* Glomerular filtration rate < 60ml/min/1.73m2 (by Chronic Kidney DIsease Epidemiology Collaboration formula)
* Known or suspected disease affecting the function of liver
* Preoperative use of strong opioids
* Patient is pregnant, cognitively disabled, under guardianship, a prisoner or in compulsory military service
* Patient will be operated by a surgeon who has done less than 100 total knee arthroplasty procedures before or by a surgeon who does not operate with Triathlon endoprosthesis
* Day of the surgery is not suitable for study (no research personnel available for 24 hours postoperative evaluation)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 402 (Actual)
Dates: Start 2016-10-03 (Actual); Primary Completion 2018-12-22 (Actual); Study Completion 2019-12-03 (Actual)

PRIMARY OUTCOMES:
Opioid consumption | 24 hours postoperative
  Cumulative intravenous oxycodone consumption By patient controlled analgesia (PCA) 24 hours postoperative.

SECONDARY OUTCOMES:
Acute postoperative pain | 24 hours postoperative
  Patient reported pain (supine at rest, with knee straight and hip in 45 degrees flexion, with knee at 45 degrees flexion and after walking 5 meters) by numerical rating scale (NRS; a whole number from 0 to10 where 0 = no pain and 10 = worst possible pain) 24 hours postoperative.
Postoperative nausea | an average of 0-3 hours and 24 hours postoperative
  Patient reported nausea by numerical rating scale (NRS; a whole number from 0 to10 where 0 = no nausea and 10 = worst possible nausea) before transferring from recovery room to surgical ward and 24 hours postoperative.
Medications given for postoperative nausea and vomiting (PONV) | an average of 2 to 3 days postoperative
  The number of medications given for PONV during postoperative hospital stay.
Chronic postoperative pain | an average of 1-2 weeks preoperative, 3 and 12 months postoperative
  Differences in Brief Pain Inventory Short Form (BPI-SF) questionnaires self-reported By patients preoperatively and 3 and 12 months postoperatively.
Predictive value of chronic pain risk index | an average of 1-2 weeks preoperative and 24 hours, 3 months and 12 months postoperative
  4 out of 5 risk factors described by Althaus et al. are asked during preoperative visit and 1 out of 5 risk factors will be assessed 24 hours postoperative. These results will be compared to results from BPI-SF questionnaires.
Knee function | an average of 1-2 weeks preoperative, 3 and 12 months postoperative
  Differences in Oxford knee score (OKS) questionnaires self-reported By patients preoperatively and 3 and 12 months postoperatively.
Self-reported quality of life | an average of 1-2 weeks preoperative, 3 and 12 months postoperative
  Differences in 15-dimensional, generic, standardized, self-administered measure of health-related quality of life (15D) questionnaires self-reported by patients preoperatively and 3 and 12 months postoperatively.
Patient satisfaction and self-reported complications | 3 and 12 months postoperative
  A patient-reported outcome measures (PROM) questionnaire made for this study including 10 questions about patient satisfaction and possible complications at 3 and 12 months postoperatively.
Times at the operation unit | from operating room to end of treatment in recovery room, an average of 3-5 hours
  Time (in minutes) spent for managing anesthesia and surgery, in the operating room and in the recovery room. Information is gathered from electrical anesthesia management program.
Need for "rescue" analgesia | From recovery room to the end of hospital stay, an average of 2-3 days
  Proportion of patients needing "rescue" analgesia in form of medications and regional anesthetic techniques outside the study protocol during the postoperative hospital stay.
Need for vasoactive medications, urine catheter and ventilatory support | intraoperative - an average of 2-3 days
  Proportion of patients needing vasoactive medications intra- or postoperatively and patients needing urine catheter or ventilatory support postoperatively.
Bleeding | 3 months to 1 day preoperative, intraoperative, 15-24 hours postoperative
  The amount of bleeding during the operation and the change in blood hemoglobin level.
Complications | 12 months postoperative
  Recorded complications derived from patient information systems up to 12 months postoperative.
Hospital length of stay | an average of 2 to 3 days up to 3 months
  Time from the start of operation to the time when patient meets the hospital discharge criteria and time when patient is actually discharged.

CONTACTS AND LOCATIONS:
Locations (1):
- Helsinki University Central Hospital, Peijas hospital, Vantaa, Finland

REFERENCES:
- [Background] Althaus A, Hinrichs-Rocker A, Chapman R, Arranz Becker O, Lefering R, Simanski C, Weber F, Moser KH, Joppich R, Trojan S, Gutzeit N, Neugebauer E. Development of a risk index for the prediction of chronic post-surgical pain. Eur J Pain. 2012 Jul;16(6):901-10. doi: 10.1002/j.1532-2149.2011.00090.x. Epub 2011 Dec 23. PMID 22337572
- [Derived] Rantasalo MT, Palanne R, Juutilainen K, Kairaluoma P, Linko R, Reponen E, Helkamaa T, Vakkuri A, Olkkola KT, Madanat R, Skants NKA. Randomised controlled study comparing general and spinal anaesthesia with and without a tourniquet on the outcomes of total knee arthroplasty: study protocol. BMJ Open. 2018 Dec 22;8(12):e025546. doi: 10.1136/bmjopen-2018-025546. PMID 30580277